CLINICAL TRIAL: NCT06966375
Title: Pilot Testing of the Worldwide Yearly Screening for Hypospadias
Brief Title: Worldwide Yearly Screening for Hypospadias
Acronym: WYSH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-0402; 2K12DK100022-06 (NIH); A539800 (Other: UW Madison); Protocol Version (Other: UW Madison)
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-08

CONDITIONS: Hypospadias
Keywords: Hypospadias Complications; Quality of Life; Patient-Reported Outcomes
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Male Participants with Repaired Hypospadias (Experimental): * 3-5 Males, age 5-10 (with parental consent and child assent)
  * 3-5 Males, age 11-15 (with parental consent and child assent)
  * 3-5 Males, age 16-20 (with parent consent, child assent until age 18)
  * 3-5 Males, age 21-65
  Interventions: Other: WYSH Web Application

INTERVENTIONS:
Other: WYSH Web Application — Worldwide Yearly Screening for Hypospadias (WYSH) Web Application

SUMMARY:
The purpose of this study is to recruit approximately 20 male participants who have a history of repaired hypospadias to test the feasibility and acceptability of the Care Planning Tool within the Worldwide Yearly Screening for Hypospadias (WYSH) Web Application.

DETAILED DESCRIPTION:
Several studies show that patients who undergo hypospadias repair report significant functional and psychosexual issues in adolescence or adulthood (in more than 50% of cases). The Care Planning tool within the Worldwide Yearly Screening for Hypospadias (WYSH) Web Application, developed using expert level consensus from a Delphi Measure including stakeholders (psychologists, urologists, endocrinologists, patients/families), is designed to support the functional and psychosexual health of male youth and adults treated for hypospadias, to support their physical and mental health after repair.

This is a pilot study of the WYSH intervention to access its feasibility and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Males who have a documented history of repaired hypospadias.
* Age groups targeted, based on recommended standards for user experience data from pilot studies:

  * 3-5 Males, age 5-10 (with parental consent and child assent)
  * 3-5 Males, age 11-15 (with parental consent and child assent)
  * 3-5 Males, age 16-20 (with parent consent, child assent until age 18)
  * 3-5 Males, age 21-65

Exclusion Criteria:

-

Ages: 5 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Participant Count to Summarize answers of the Care Planning Tool | Baseline, 3 weeks, 3 months
  The Care Planning Tool within the Worldwide Yearly Screening for Hypospadias (WYSH) Application is a survey containing forty-eight questions regarding possible complications for participating patients (Subsections of penile function, voiding, sexual health, social functioning, psychological health, and doctor-patient communication). These questions will be completed by patients using a five point scale - "Never," "Rarely," "Sometimes," "Often," and "Always" - to populate a Care Plan highlighting areas of concern (with a threshold of two or more metrics above a "Sometimes" response).
Acceptability: User Centered Metrics | Baseline, 3 weeks, 3 months
  Participating patients will complete a survey regarding the System Usability to determine ease of functionality throughout the application. This survey contains a scale for participants to graph their response from "Very Difficult" to "Very Easy" following the eleven questions of task completion. Additionally, there is a space provided for open-ended feedback.
Acceptability: Cognitive Debriefing Measures | Baseline, 3 weeks, 3 months
  A team from the Wisconsin Surgical Outcomes Research Program (WiSOR) will complete a Cognitive Debriefing Interview with participating patients to assist in determining validation and comprehension. This interview consists of seven open-ended questions regarding participants' thought processes to provide an insight into areas of improvement for the application. Answers will be coded and themes summarized by participant count.
Feasibility: System Usability Testing | Baseline, 3 weeks, 3 months
  The Center for User Experience will conduct masked System Usability Testing to provide user-based information on how to improve the online experience for young males and their caregivers and adult males. Usability will be assessed with a level of success rating from "Failure," "Success with a major issue," "Success with a minor issue," and "Complete Success," where minor or major issues and time taken are observed as the participating patient is completing the System Usability Scale.

SECONDARY OUTCOMES:
Provider Acceptability: Usability Scale | Data collected after participating patient completes questionnaire, up to approximately 3 months.
  Participating UW Clinicians will rate the recommendations received in each care plan from patients in a separate usability scale (Provider Acceptability) to improve the ability for continuity of care. Providers will complete a survey of questions surrounding format, output, and utility from "Strongly Disagree" to "Strongly Agree." Additionally, there is a space provided for feedback.

CONTACTS AND LOCATIONS:
Overall Officials: Vinaya Bhatia, MD, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- UW School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during pilot testing, after deidentification, will be accessible in the form of text, tables, publications, figures, etc. to disseminate efficacy of the Care Planning tool within the application.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Deidentified individual personal data and supporting information will be made available immediately after publication.